CLINICAL TRIAL: NCT01030627
Title: Treatment Approaches to Preeclampsia
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Gynuity Health Projects (Other)
Collaborators: Daga Memorial Women's Hospital, Nagpur, India (Other); Matra Sewa Sangh, Nagpur, India (Unknown); University of Washington (Other)
Responsible Party: Beverly Winikoff, Gynuity Health Projects
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 4.2.2
Record Dates: First submitted 2009-12-10; First posted 2009-12-11 (Estimated); Last update posted 2011-08-11 (Estimated); Status verified 2011-08

CONDITIONS: Preeclampsia
Keywords: Eclampsia; Preeclampsia; Magnesium sulfate
MeSH Terms: conditions — Pre-Eclampsia; Eclampsia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: Springfusor infusion pump — Women will receive a loading dose and maintenance therapy using an IV infusion administered by the Springfusor® pump. Women will receive a 8 mL loading dose containing 4g magnesium sulfate heptahydrate (MgSO4*7H2O) 50% solution, which is approximately 2 mmoL magnesium/mL. The loading dose of 8mL with 4 g MgSO4 will be administered using the Springfusor® pump. The administration of the loading dose will be immediately followed by a maintenance infusion. The maintenance dose of 4 g (8 cc, 50% MgSO4) will be administered with the Springfusor® pump continuously over four hours. The pump will be started immediately after the initial bolus and the 4g dose repeated (and syringe replaced) every four hours. Maintenance therapy will be administered for at least 24h. Treatment will be discontinued when clinically indicated. Drug administration will be initiated at the sites and, when necessary, the patient will be transferred, with the Springfusor pump in situ, to the local referral site.

SUMMARY:
This pilot study will document the efficacy and acceptability of administration of magnesium sulfate with the Springfusor pump for patients and staff at two sites where treatment or preeclampsia with magnesium sulfate is limited or not available. Currently, both sites refer patients to tertiary care facilities for further treatment.

DETAILED DESCRIPTION:
Women diagnosed with preeclampsia that the clinic care team deem would benefit from treatment with magnesium sulfate will be given the option of participating in the study. Those who choose to take part in the study and meet study inclusion and exclusion criteria will receive full information about the study and be required to give their written or signed informed consent.

Women agreeing to participate in the study will receive a loading dose and maintenance therapy using an IV infusion administered by the Springfusor® pump. Women will receive a 8 mL loading dose containing 4g magnesium sulfate heptahydrate (MgSO4*7H2O) 50% solution, which is approximately 2 mmoL magnesium/mL. The loading dose of 8mL with 4 g MgSO4 will be administered using the Springfusor® pump. The administration of the loading dose will be immediately followed by a maintenance infusion. The maintenance dose of 4 g (8 cc, 50% MgSO4) will be administered with the Springfusor® pump continuously over four hours. Clinical monitoring will occur once every hour during the treatment period. Clinical monitoring will occur throughout the treatment, with reflexes, urine output and respiration to be checked at least every hour (or, if more frequent, as per standard practice at the study site). The pump will be checked at each monitoring visit. Prior to discharge from the study, patients will be asked to assess their opinions about the acceptability and ease of use of the mode of administration. All requests or inquiries about termination of treatment will be recorded.

ELIGIBILITY:
Inclusion Criteria:

* Exhibit systolic blood pressure > 140mm Hg OR a diastolic pressure > 100 mm Hg
* Exhibit proteinuria > 1+
* Have not given birth, or be 24h or less postpartum
* Exhibit urine output >100 ml or more during the previous 4h or greater than 25 mL/h
* Agree to comply with study procedures
* Be > 18 years of age
* Give informed consent for study participation

Exclusion Criteria:

* Eclamptic or seizing at the time of enrollment
* Received magnesium sulfate therapy 24h prior to study enrollment

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 85 (Actual)
Dates: Start 2009-10; Primary Completion 2010-04 (Actual); Study Completion 2010-04 (Actual)

PRIMARY OUTCOMES:
Completion of full course of treatment | 24 hours

CONTACTS AND LOCATIONS:
Overall Officials: Beverly Winikoff, MD, Principal Investigator — Gynuity Health Projects; Thomas Easterling, MD, Principal Investigator — University of Washington
Locations (2):
- India (2):
  - Daga Memorial Women's Hospital, Nagpur, Maharashtra
  - Matra Sewa Sangh, Nagpur

REFERENCES:
- See also: Gynuity Health Projects — http://www.gynuity.org